CLINICAL TRIAL: NCT05027659
Title: The Effects of Virtual Reality Glasses on Vital Signs and Anxiety in Patients Undergoing Colonoscopy: A Randomized Controlled Trial
Brief Title: The Effects of Virtual Reality Glasses on Vital Signs and Anxiety in Patients Undergoing Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esra DOĞAN YILMAZ, RN, MSc (Other)
Responsible Party: Sponsor-Investigator, Esra DOĞAN YILMAZ, RN, MSc, Research Assistant, Kırıkkale University
Organization: Kırıkkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EYILMAZ-experimental study
Record Dates: First submitted 2021-07-15; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Vital Signs; Anxiety; Colonoscopy
Keywords: Anxiety; colonoscopy; pain; virtual reality glasses; vital signs
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The data of the study were entered by a person other than the researcher. Statistical analysis was performed by a person other than the researcher. In the study, virtual reality glasses were worn on the participants of experimental group. For this reason, blinding could not be done for the participants. The researcher herself collected all data because the hospital restricted traffic in and out of the unit due to the pandemic. Therefore, the evaluator was not blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): This study was carried out with two groups. Virtual reality glasses were used for the intervention group.
  Interventions: Other: virtual reality glasses
- control (No Intervention): No application was made to the control group, standard procedure was followed.

INTERVENTIONS:
Other: virtual reality glasses — Virtual reality (VR) glasses have a detachable screen frame compatible with smartphones. A VR headset has earphones and sensors that track the user's head movements, giving them the impression that they are moving around in a virtual environment. The investigators used a smartphone and VR glasses to perform the intervention. They connected the phone to the VR headset via a 360 degree VR video app. Experimental participants wore the VR glasses and watched a 360 degree VR video of nature scenes with ambiance music during colonoscopy. They put on the VR glasses right before the procedure and took them off right afterward.
  Arms: intervention

SUMMARY:
The present study was conducted with 44 patients who applied to the Endoscopy Unit of a university hospital for sedation-free colonoscopy between January 2, 2020 and September 28, 2020, met the inclusion criteria and agreed to participate in the study. The patients were homogeneously divided into experimental (n=22) and control (n=22) groups based on their gender and history of colonoscopy. The patients in the experimental group watched a 360 degree virtual reailty (VR) video with atmospheric background music over images and sounds of nature through virtual reality glasses while no application was performed for the patients in the control group during the procedure. The "Demographic Information Form", "Trait Anxiety Scale", "Visual Analog Scale-Pain", "Visual Analog Scale-Anxiety", "Vital Signs Monitoring Chart" and "Satisfaction Evaluation on the Virtual Reality Glasses Application" forms were used in the data collection phase. For the study, an ethics committee approval was obtained in addition to written consent by the institutions and patients. Numbers, percentages, the Chi-square test, the Wilcoxon test and the Mann-Whitney U test were used for data analysis.

DETAILED DESCRIPTION:
Aims: This study investigated the effect of VR glasses on vital signs and anxiety in patients undergoing colonoscopy. The research questions are as follows:

* Wearing VR glasses during colonoscopy affects at least one vital sign.
* Wearing VR glasses during colonoscopy affects anxiety. Study design and setting: This study adopted a randomized controlled experimental design. The study population consisted of all patients (N=82) who had a colonoscopy without sedation between January 2, 2020, and September 28, 2020, at the endoscopy unit of a training and research hospital in Kırıkkale, Turkey. Patients were randomized into experimental and control groups before the procedure.

Group 1 (experimental): Virtual reality glasses have a detachable screen frame compatible with smartphones. A VR headset has earphones and sensors that track the user's head movements, giving them the impression that they are moving around in a virtual environment (Arane et al., 2017; Indovina et al., 2018). The investigators used a smartphone and VR glasses to perform the intervention. They connected the phone to the VR headset via a 360o VR video app. Experimental participants wore the VR glasses and watched a 360o VR video of nature scenes with ambiance music during colonoscopy. They put on the VR glasses right before the procedure and took them off right afterward.

Each control group participant (Group 2) underwent the standard procedure.

Sample size calculation: The sample consisted of 44 participants divided into experimental (n=22) and control (n=22). A post-power analysis was conducted on Visual Analog Scale-Pain (VAS-P) scores due to the pandemic. The results showed that the sample was large enough to detect significant differences (effect size = 1.31; type I margin of error (α) = 0.05; test power (1-β) = 0.98).

Randomization: Simple stratified randomization was used for homogeneity.Participants were assigned to the groups based on their gender and colonoscopy history.For each patient randomly assigned to a group (drawing lots), another patient with the same gender and colonoscopy history was included in the other group. For example, the investigators wrote down "experimental" and "control" on pieces of paper for a female participant scheduled for a colonoscopy for the first time and put them in a bag. Then, they asked the nurse in charge to pull one of the pieces of paper out of the bag. In this way, that participant was assigned to the group written on the piece of paper. Afterward, the investigators assigned another patient with the same gender and colonoscopy history to the other group. The nurse pulled a new piece of paper out of the bag for a patient with a different gender and colonoscopy history. The investigatorsassigned that patient to the corresponding group. They followed the same procedure for all groups (Woman-first time colonoscopy; Woman- colonoscopy before; Man-first time colonoscopy; Man- colonoscopy before) to achieve homogenous groups.

Research shows that gender and colonoscopy history affect pain and anxiety during colonoscopy. Therefore, the investigators used the same parameters to randomize participants into the groups, which were similar in terms of gender and colonoscopy history.

Data collection tools: Data were collected using a demographic characteristics questionnaire and the Visual Analog Scale-Anxiety (VAS-A). Vital signs (Blood pressure, pulse rate, and SpO2) were also measured using a monitor. The respiratory rate was measured by the researcher. The pain was assessed using the Visual Analog Scale-Pain (VAS-P). A five-point scale ("very satisfied,""satisfied,""undecided,""dissatisfied," and "very dissatisfied") was used to determine how satisfied participants were with wearing the VR glasses during the procedure.

Research Implementation: Patients were informed about the research purpose and procedure, and consent was obtained from those who agreed to participate. All participants filled out the demographic characteristics questionnaire, VAS-P, and VAS-A, and their vital signs were measured before colonoscopy. The experimental group participants wore the VR glasses and watched a 360 degree VR video of nature scenes with ambiance music during colonoscopy. The control group participants underwent the standard procedure. All participants filled out the VAS-P and VAS-A, and their vital signs were measured after the procedure. How satisfied the experimental group participants were with the VR application was also assessed after the procedure.

Ethical Consideration: The study was approved by an ethics committee (Date: 31.07.2019 & No:44). Permission was obtained from the hospital (Date: 07.08.2019 & No: 28955). Patients were informed about the research purpose, procedure, and confidentiality prior to participation and that they could withdraw from the study at any time without any monetary concessions. Written consent was obtained from those who agreed to participate. Permission was obtained from the developer of the 360 degree VR video.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary
* Scheduled for a colonoscopy without sedation
* Aged 18 to 79 years
* No perception, hearing, and vision impairment that interferes with communication
* Not wearing glasses
* No psychiatric disorder
* No migraine, vertigo, active nausea, vomiting, headache, etc.

Exclusion Criteria:

* no Voluntary
* Scheduled for a colonoscopy with sedation
* not been Aged 18 to 79 years
* participants have been perception, hearing, and vision impairment that interferes with communication
* wearing glasses
* participants have psychiatric disorder
* participants have migraine, vertigo, active nausea, vomiting, headache, etc.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Research shows that gender affect pain and anxiety during colonoscopy. Therefore, we randomized participants into the groups, which were similar in terms of gender.
Enrollment: 44 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
blood pressure | Change in systolic blood pressure during colonoscopy, an average of 20 minutes
  mmHg. higher scores mean a worse
pulse rate (heart rate) | Change in pulse rate during colonoscopy, an average of 20 minutes
  beats per minute. higher scores mean a worse
respiratory rate | Change in respiratory rate during colonoscopy, an average of 20 minutes
  respiratory rate per minute. higher scores mean a worse
peripheral oxygen saturation (SpO2) | Change in peripheral oxygen saturation during colonoscopy, an average of 20 minutes
  Approaching 100% is considered positive. higher scores mean a better
Pain score | Change in pain score during colonoscopy, an average of 20 minutes
  Visual Analog Scale-Pain (VAS-P), which is a 10cm long line with anchor statements "0=no pain" at the left-most end and "10=unbearable pain" at the right-most end. minimum=0, maximum=10; higher scores mean a worse and lower scores mean a better
Anxiety score | Change in anxiety score during colonoscopy, an average of 20 minutes
  Visual Analog Scale-Anxiety (VAS-A), which is a 10 cm long horizontal line with anchor statements "0=no anxiety at all" at the left-most end and "10=worst anxiety imaginable" at the right-most end. minimum=0, maximum=10; higher scores mean a worse and lower scores mean a better

CONTACTS AND LOCATIONS:
Overall Officials: Esra DOĞAN YILMAZ RN, PhD, Research Assistant, Principal Investigator — Kırıkkale University
Locations (1):
- Kirikkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The confidentiality of the data used in the study will be protected.

REFERENCES:
- [Derived] Dogan Yilmaz E, Unlusoy Dincer N. The Effects of Virtual Reality Glasses on Vital Signs and Anxiety in Patients Undergoing Colonoscopy: A Randomized Controlled Trial. Gastroenterol Nurs. 2023 Jul-Aug 01;46(4):318-328. doi: 10.1097/SGA.0000000000000733. Epub 2023 Jun 5. PMID 37278621